CLINICAL TRIAL: NCT05815602
Title: Multicenter Randomized Controlled Clinical Trial Comparing Ebastine and Mebeverine as Treatment of Irritable Bowel Syndrome
Brief Title: Ebastine Versus Mebeverine in IBS Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guy Boeckxstaens (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor-Investigator, Guy Boeckxstaens, prof. dr., KU Leuven
Organization: KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S67029
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: IBS - Irritable Bowel Syndrome; IBS
Keywords: ebastine; duspatalin; IBS; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — ebastine; mebeverine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ebastine verum and duspatalin placebo (Experimental)
  Interventions: Drug: Ebastine
- Duspatalin verum and ebastine placebo (Active Comparator)
  Interventions: Drug: Duspatalin

INTERVENTIONS:
Drug: Ebastine — Randomized subjects will administer 4 pills of study medication per day during 12 weeks.
  Daily administration schedule consists of taking 2 pills in the morning (1 verum, and 1 placebo). In the evening, subjects will take a second dose of both verum and placebo.
  Arms: Ebastine verum and duspatalin placebo
Drug: Duspatalin — Randomized subjects will administer 4 pills of study medication per day during 12 weeks.
  Daily administration schedule consists of taking 2 pills in the morning (1 verum, and 1 placebo). In the evening, subjects will take a second dose of both verum and placebo.
  Arms: Duspatalin verum and ebastine placebo

SUMMARY:
Multicenter randomized controlled clinical trial comparing ebastine and mebeverine as treatment of irritable bowel syndrome

Trial rationale

1. To perform a randomized superiority trial comparing the clinical efficacy of ebastine and mebeverine
2. To evaluate the impact of treatment with ebastine compared to mebeverine on quality of life and quality-adjusted life years

Primary objective To provide further evidence of the superiority of histamine 1 receptor antagonism as novel treatment for patients with non-constipated IBS, as compared to mebeverine, one of the spasmolytics currently used as first line treatment of IBS.

Secondary objective(s) To provide evidence that the histamine 1 receptor antagonist ebastine is more effective in reducing abdominal pain compared to the commonly used antispasmodic mebeverine

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. Patients fulfilling the Rome IV criteria for non-constipated IBS (IBS-C subtypes will be excluded)
3. No organic cause that can explain the presenting symptoms (exclusion of coeliac disease (blood), lactose intolerance (breath test), inflammatory bowel disease and giardiasis (stool)
4. Patients with lactose intolerance can be included if no improvement on lactose free diet during 6 weeks
5. Age 18-65

Exclusion Criteria:

1. History of coeliac disease, food allergy, giardiasis, inflammatory bowel disease, infectious gastroenteritis, motility disorder, serious liver kidney cardiac or pulmonary disease, known cardiac rhythm disorders, insuline-dependent diabetes, psychiatric diseases
2. Pregnancy, breast feeding
3. Medication: the use of antidepressants or antipsychotics, anti-allergic medication or drugs affecting gastrointestinal motility / visceral sensitivity (anti-cholinergics, antispasmodics, 5-HT3 antagonists, 5-HT4 agonists, loperamide, codeine, laxatives, analgesics: only paracetamol is allowed as analgetic, other analgesics are forbidden.), CYP3A4-inducing and inhibiting drugs. Potent inhibitors of CYP3A4 include clarithromycin, erythromycin, diltiazem, itraconazole, ketoconazole, ritonavir, verapamil, goldenseal and grapefruit. Inducers of CYP3A4 include phenobarbital, phenytoin, rifampicin, St. John's Wort and glucocorticoids.
4. Symptoms started following abdominal surgery
5. IBS constipation dominant (IBS-C)
6. Hypersensitivity to the active substance or to any of the excipients listed in section 6.1 of the SmPC of the respective medicinal products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Response to Abdominal Pain Intensity | 12 weeks of study medication administration
  The primary endpoint is defined as Clinical Response to Abdominal Pain Intensity and Global Relief of Symptoms. A clinical responder is defined to be a Weekly Responder for both Abdominal Pain Intensity and Global Relief of Symptoms for at least 3 out of the 6 last weeks of treatment.
  Abdominal Pain Intensity is assessed daily by the subject during the 14 days prior to (run-in) and following (run-out) randomization and for 12 weeks during treatment, using a 10-point scale. For each week during and following treatment, an average pain score is calculated. Then %change from the mean baseline will be calculated. An Abdominal Pain Intensity Weekly Responder is defined as a subject who had a decrease of >=30% compared with baseline.
Clinical Response to Global Relief of Symptoms | 12 weeks of study medication administration
  Global Relief of Symptoms is assessed on a weekly basis using a 7-point scale for 12 weeks during treatment and run-out: a Weekly Responder is defined if he has total or obvious relief of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Boeckxstaens, prof. dr., Principal Investigator — KU Leuven
Locations (5):
- Belgium (5):
  - AZ St-Maarten, Mechelen, Antwerpen
  - UZLeuven, Leuven, Vlaams-Brabant
  - AZ St-Lucas, Bruges, West-Vlaanderen
  - GZA, Antwerp
  - UZA, Antwerp

IPD SHARING:
Plan to Share IPD: No